CLINICAL TRIAL: NCT04502771
Title: Therapeutic Drug Monitoring of Antifungals in Patients From Intensive Care Units: a Retrospective Study
Brief Title: Therapeutic Drug Monitoring of Antifungals in Intensive Care Units
Acronym: Fungi-up
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2020_003
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Intensive Care Unit Patients
Keywords: Fluconazole; Voriconazole; Posaconazole; Caspofungin; Therapeutic drug monitoring; Blood concentration; Under-dosing; Over-dosing; Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Antifungal treatment: Patients receiving antifungal treatment during their stay in Intensive Care Unit
  Interventions: Drug: Antifungal treatment

INTERVENTIONS:
Drug: Antifungal treatment — Treatment by fluconazole, voriconazole,posaconazole or caspofungin during the patient stay in Intensive Care Unit

SUMMARY:
Antifungals under- and over-dosing are frequently deplored in patients treated with antifungals and receiving recommended doses, mostly in critically-ill patients. This situation is well-described for antifungals from the azoles class mostly in patients with liver dysfunction or having concomitant drugs that may interact with azoles. This situation is less-described using echinocandins, although recent studies reported caspofungin underdosing for critically-ill patients. Considering that antifungals under-dosing was demonstrated to be associated with an increase in mortality, it is of utmost importance to analyse the relevance of therapeutic drug monitoring (TDM) for patients admitted in intensive care units (ICU). This will help to identify which patients are the more prone to antifungal under or over-dosing. Indeed, antifungals under-dosing may favour the development of clinical resistance to antifungals and increase mortality, whereas over-dosing may result in adverse events that may lead to treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who received antifungals including fluconazole, voriconazole, posaconazole, or caspofungin, during their ICU stay and had a Therapeutic Drug Monitoring (TDM)

Exclusion Criteria:

* Patients without antifungal treatment
* Patients who received an antifungal combination
* Pediatric patients
* Patients who were not admitted in ICU
* Patients who did not have a TDM

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received antifungals during their ICU stay and had a TDM
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Antifungal blood concentration of patients admitted in intensive care units | Day 5 after antifungal initiation

SECONDARY OUTCOMES:
Adverse event | Day 30 after antifungal initiation
  Impact of antifungal blood concentration on occurrence of adverse events and mycological failure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Croix-Rousse Hospital, Lyon, France